CLINICAL TRIAL: NCT02819648
Title: The Effect of Preoperative Oral Administration of Prednisolone on Postoperative Pain in Patients With Symptomatic Irreversible Pulpitis: A Single Center Randomized Controlled Trial
Brief Title: Oral Glucocorticoids Effect on Post Endodontic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Elkhadem, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCRCT1
Record Dates: First submitted 2016-06-24; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Pulpitis
Keywords: symptomatic; irreversible
MeSH Terms: conditions — Pulpitis | interventions — Prednisolone; Glucocorticoids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisolone (Experimental): 40 mg prednisolone (two tablets Prednisolone 20 mg, Aventis Intercontinental, Paris, France); administered 30 minutes before endodontic treatment
  Interventions: Drug: Prednisolone
- Control (Placebo Comparator): Milk tablet administered 30 minutes before endodontic treatment
  Interventions: Other: Control

INTERVENTIONS:
Drug: Prednisolone — 40 mg prednisolone (two tablets Prednisolone 20 mg, Aventis Intercontinental, Paris, France)
  Other Names: Glucocorticoid
  Arms: Prednisolone
Other: Control — Milk Tablet
  Other Names: Placebo
  Arms: Control

SUMMARY:
The aim of this single-center randomized, double-blind, placebo-controlled clinical trial is to assess the effect of preoperative, single, oral dose of prednisolone on postoperative pain and medication intake in patients with symptomatic, irreversible pulpitis in mandibular molars.

DETAILED DESCRIPTION:
Patients receive 40 mg prednisolone (two tablets Prednisolone 20 mg, Aventis Intercontinental, Paris, France); and group B (Control), where patients received two placebo tablets. All patients receive the assigned premedication 30 minutes before the administration of local anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients, aged between 18-35 years, with mandibular molars with symptomatic irreversible pulpitis, radiographically-normal periapical area and no pain on biting or percussion.

Exclusion Criteria:

* Pregnant patients, patients with any known sensitivity or adverse reactions to any of the medications or materials used in this study, those who had used any analgesic medication during the preceding 6 hours before the treatment, those with unrestorable teeth or teeth with severe periodontal disease. Patients with active sites of pathosis in the area of injection were, also, excluded.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2012-06; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Degree of postoperative pain using a visual analogue scale (VAS) | 24 hours
  Measured using visual analogue scale (VAS). It is a 10 points scale from 0 to 10, where zero expresses no pain and 10 expresses severe pain

SECONDARY OUTCOMES:
Intake of fake analgesic (sham) following endodontic treatment (Binary outcome) | 24 hours
  This is a binary outcome (Intake/No intake). Each patient is given one milk tablet (sham) and instructed to use it only if patient feels post-operative pain. The aim of using a fake analgesic is to minimize the use of true analgesic which might mask the post-operative pain scoring in the first 24 hours.
Intake of true analgesic following endodontic treatment (Binary outcome) | 24 h
  This is a binary outcome (Intake/No intake). Each patient is given one tablet of analgesic (Diclofenac Potassium 50 mg, Novartis Pharma, Ontario, Canada). Patient is instructed to use it only if patient post-operative pain exists 2 hours following sham (fake analgesic) intake.

CONTACTS AND LOCATIONS:
Overall Officials: Suzan Wanees, PhD, Principal Investigator — Cairo Univeristy
Locations (1):
- Faculty of Oral & Dental Medicine, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Through journal publication

REFERENCES:
- [Result] Jalalzadeh SM, Mamavi A, Shahriari S, Santos FA, Pochapski MT. Effect of pretreatment prednisolone on postendodontic pain: a double-blind parallel-randomized clinical trial. J Endod. 2010 Jun;36(6):978-81. doi: 10.1016/j.joen.2010.03.015. Epub 2010 Apr 24. PMID 20478449